CLINICAL TRIAL: NCT06341647
Title: A Multicenter, Open-label, Phase 1 Clinical Trial to Evaluate the Safety and Anti-Tumor Activity of AB-201 in Subjects With Advanced Human Epidermal Growth Factor Receptor 2 Positive(HER2+) Solid Tumors
Brief Title: Phase 1 Clinical Trial to Evaluate the Safety and Anti-Tumor Activity of AB-201
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Determined that enrollment would be limited due to the change in care setting.
Sponsor: GC Cell Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AB-201-01; 103300 (HREC 233/23) (Other: TGA (Australia))
Record Dates: First submitted 2024-03-14; First posted 2024-04-02 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: * Safety: incidence and severity of AE and SAE [Time Frame: From the time of consent through End of Study (up to 18 months per patient)]
  * Determination of Recommended Phase 2 Dose (RP2D)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1a Dose Escalation (Experimental): * Dose Escalation of AB-201 in advanced metastatic breast cancer, gastric or gastroesophageal junction adenocarcinoma with HER2 overexpression
  * Interventions:
    * Drug: AB-201
    * Drug: Cyclophosphamide
    * Drug: Fludarabine
  Interventions: Drug: AB-201; Drug: Cyclophosphamide; Drug: Fludarabine
- Phase 1b Dose Expansion (Experimental): * Dose Confirmation of AB-201 in advanced metastatic breast cancer, gastric or gastroesophageal junction adenocarcinoma with HER2 overexpression
  * Interventions:
    * Drug: AB-201
    * Drug: Cyclophosphamide
    * Drug: Fludarabine
  Interventions: Drug: AB-201; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: AB-201 — NK Cell Therapy
Drug: Cyclophosphamide — Lymphodepleting chemotherapy
Drug: Fludarabine — Lymphodepleting chemotherapy

SUMMARY:
This clinical trial will enroll subjects with HER2+ solid tumors and is conducted in two phases, which are phase 1a and phase 1b. The primary objective of phase 1 is to determine the safety and tolerability of AB-201 in subjects with advanced HER2+ solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter study designed to evaluate the safety, tolerability, and efficacy of AB-201 in subjects with advanced HER2+ solid tumors (specifically, breast and gastric/GEJ cancers).

The Phase 1 will be conducted in two parts, an initial dose escalation stage followed by a dose expansion stage.

Study participation for each subject begins with up to 28 days (1 month) of screening following written informed consent, then lymphodepletion treatment, followed by AB-201. Up to 3 doses of AB-201 may be administered. All subjects will be monitored for a total duration of 18 months of follow up from the first dose administration of AB-201.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0 to 1.
* Histologically confirmed HER2 expressed breast or gastric/GEJ cancer IHC ≥ 2+ within 6 months prior to study entry.
* Confirmed diagnosis of an advanced/unresectable or metastatic HER2+ breast or gastric/GEJ cancer that is refractory to, or intolerable of standard treatment, or for which no standard treatment is available.
* Must have received prior cancer therapy: Subjects with breast cancer must have received ≥ 3 prior systemic therapies; subjects with gastric/GEJ cancer must have received ≥ 2 prior systemic therapy(ies); subjects with IHC 3+ or IHC 2+/ISH+ cancers must have received previous treatment with a HER2-targeting therapy.

Exclusion Criteria:

* Known past or current malignancy other than inclusion diagnosis.
* Known clinically significant cardiac disease.
* Active central nervous system (CNS) metastases, or involvement of the CNS, unless there is a history of at least 3 months of sustained remission.
* Unresolved toxicities from prior anticancer therapy.
* Ongoing uncontrolled systemic infections requiring antibiotic, anti-fungal, or anti-viral therapy.
* History of sensitivity or intolerance to cyclophosphamide or fludarabine.
* Currently Pregnant or lactating
* Severe disease progression or health deterioration within 2 weeks prior to lymphodepletion regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, seriousness, and dose relationship of Adverse Events [Safety & Tolerability] | up to 18 months per patient
  Adverse events and laboratory abnormalities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Determination of Recommended Phase 2 Dose (RP2D) | up to 18 months per patient
  Assessment of Dose-Limiting Toxicities(DLTs), pharmacokinetics (PK), safety, and objective response rate (ORR) per the Response Evaluation Criteria for Solid Tumors (RECIST) v1.1 in subjects with HER2+ breast cancer and gastric/GEJ cancer.
  PK: Monitor persistence of AB-201 in subjects samples collected prior to and following AB-201 administration.

SECONDARY OUTCOMES:
To determine the preliminary efficacy, by the objective response rate (ORR) per the Response Evaluation Criteria for Solid Tumors (RECIST) v1.1, of AB-201 in subjects with advanced HER2+ solid tumors | up to 18 months per patient
  The proportion of subjects who experienced an PR or CR, as assessed by investigators per RECIST v1.1.

IPD SHARING:
Plan to Share IPD: No